CLINICAL TRIAL: NCT06828614
Title: Evaluation of the Barriers to Therapeutic Exercise Perceived by People With Breast Cancer Who Are Undergoing Chemotherapy in an Observational Study
Brief Title: Barriers to Therapeutic Exercise in Breast Cancer Patients Before, During, and After Chemotherapy
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, SARA CORTES AMADOR, Assistant Professor of Physiotherapy, University of Valencia
Other Study IDs: UV-INV_ETICA-3253850
Record Dates: First submitted 2025-02-04; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Chemotherapy; Barriers to exercise; Physical activity; Fatigue
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Fatigue | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-chemotherapy: Group 1 will include patients diagnosed with breast cancer who are scheduled to start chemotherapy treatment.
  Interventions: Drug: Chemotherapy
- During chemotherapy: Group 2 will include patients with breast cancer who at the time of the study are receiving chemotherapy treatment.
  Interventions: Drug: Chemotherapy
- Post-chemotherapy: Group 3 will include patients with breast cancer who have completed chemotherapy treatment 6 months or more ago.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — The present approved ethics committee includes the conduct of two studies. In the first one, a cross-sectional study, breast cancer patients will be distributed in the study groups according to the moment of their chemotherapy treatment (group 1: pre-chemotherapy, group 2: during chemotherapy, group 3: post-chemotherapy). Each patient will undergo a single evaluation session, which will include the variables detailed in the following section.
  In the second, a longitudinal study, patients from the previous study in group 1 (pre-chemotherapy) will be followed up. Patients will receive three assessments of the variables detailed in the following section: 1) during the time prior to the start of chemotherapy (assessment that will coincide with study 1), 2) assessment during chemotherapy treatment and, 3) assessment after the end of chemotherapy treatment.

SUMMARY:
Cancer is one of the leading causes of mortality. First-choice cancer treatments, such as chemotherapy, have increased the survival of people with cancer, although they are not without adverse effects such as cardiotoxicity, fatigue, nausea, mental health problems or musculoskeletal disorders.

Therapeutic exercise is a safe and effective intervention that has shown positive results in the oncology population when implemented as an adjuvant to chemotherapy, during or after chemotherapy. Exercise improves cardiorespiratory capacity, fatigue, strength, anxiety, depressive symptoms and quality of life, among others, in cancer patients.

In the implementation of therapeutic exercise in the oncologic population undergoing chemotherapy treatment, it is necessary to take into account possible barriers related to the perception of therapeutic exercise, as well as the side effects derived from chemotherapy. It is necessary to know the barriers to the implementation of exercise in order to address them and favor patients' adherence to exercise programs.

The objective is to identify the barriers (physical, contextual and emotional) that may influence people with breast cancer who are in the pre-, concurrent or post-treatment phase, respectively, of chemotherapy treatment for the implementation of therapeutic exercise.

The study participants (n=111) will be distributed in the study groups according to the moment of chemotherapy treatment they are in (1: pre-chemotherapy, 2: during chemotherapy, 3: post-chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age with a diagnosis of breast cancer, stages I to IIIa.
* The sample will be distributed to three groups according to the time of treatment in which the patients are: a) patients diagnosed with breast cancer scheduled to start chemotherapy treatment, b) patients who at the time of the study are receiving chemotherapy and c) patients who have completed chemotherapy treatment 6 months ago or more.

Exclusion Criteria:

* Women with breast cancer relapse and/or other types of cancer.
* Patients who are receiving hormonal therapy at the time of evaluation.
* Patients presenting metastatic processes or any other relevant disease.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women over 18 years of age diagnosed with breast cancer, stages I to IIIa. The patients in the sample must be in one of the following conditions: a) patients diagnosed with breast cancer with scheduled initiation of chemotherapy treatment, b) patients who at the time of the study are receiving chemotherapy and c) patients who have completed chemotherapy treatment 6 months or more ago.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Cancer-related fatigue | Day 1
  It will be evaluated with the Spanish version of the self-reported Piper Fatigue Scale. It presents 22 items and includes four dimensions related to subjective fatigue (behavioral, affective, sensory and cognitive). Scores are between 0 and 10, the higher the total score the greater the disability (0 = no fatigue, 1-3 = mild fatigue, 4-6 = moderate fatigue, 7-10 = severe fatigue).

SECONDARY OUTCOMES:
Body composition | Day 1
  It will be evaluated by means of a scale (TANITA BC-351, Japan). It uses the different impedances of the conductive and isolated parts of the body, allowing to calculate the weight (Kq). Weight and height will be combined to report BMI in kg/m^2)
Muscle strength | Day 1
  The hand grip strength test will be evaluated with a digital dynamometer (Jamar Plus+ digital hand dynamometer (Patterson Medical, Sammons Preston, Bolingbrook, IL, USA)). The patient will be placed in a seated position with the shoulder in adduction and neutral rotation, the elbow flexed at 90º and the forearm and wrist in neutral position. The maximum grip strength will be measured alternately three times on each arm, and the mean of the three measurements will be recorded.
Upper limb function | Day 1.
  It will be evaluated using the Disability of Arm, Shoulder and Hand (DASH) questionnaire. It is a scale of 30 items, of which 21 refer to the degree of difficulty in performing physical activities, 5 refer to the severity of some pain symptoms and 5 refer to other activities. The score ranges from 0 to 100 points, the higher the score the greater the disability.
Functional capacity | Day 1.
  It will be assessed by the 6-minute walk test (6MWT) on a treadmill. It determines the maximum distance a person can walk in 6 minutes. It will also include the 30 sec Sit to Stand test, which evaluates how many times the patient is able to stand and sit in a chair, with arms crossed over the chest, for 30 seconds.
Physical activity | Day 1
  This will be recorded by means of the International Physical Activity Questionnaire (IPAQ), which will allow patients to be divided according to their level of physical activity as high, moderate and low or inactive. Information on physical activity will also be collected by means of a physical activity diary, in which each patient will record the last seven days of physical activity, type of activity, intensity, duration and perceived level of fatigue.
Self-efficacy for physical activity | Day 1
  The Self-Efficacy for Physical Activity Scale (EAF) will be used, which addresses patients' beliefs about their own abilities to perform physical activities. It allows the identification of barriers and limitations that prevent the patient from engaging in regular physical activity. It presents three domains (programmed physical exercise, physical activity in daily activities and walking), which include 39 items, scored from 0 to 10, with a higher score indicating a greater capacity to perform physical activity.
Leisure time physical activity | Day 1
  This will be assessed using the abbreviated version of the Minnesota Leisure Time Physical Activity Questionnaire (VREM). It is composed of 5 items, asking about the period of a typical week in which participants perform routine household activities, as well as activities performed during the last month (e.g. walking, stair climbing, sports, dancing etc.). Gastro-energy in METs/min is calculated and the patient is classified from sedentary to very active.
Physical fitness | Day 1
  The Spanish version of the International Fitness Scale (IFIS) will be used, which measures general physical confidence, cardiorespiratory confidence, muscular strength, speed/agility and flexibility in comparison with the fitness level of a friend. It is scored on a Likert scale from very poor to very good.
Quality of life (EORT QLQ-BR23) | Day 1
  It will be assessed using the Breast Specific Quality of Life Questionnaire by the European Organisation for Research and Treatment of Breast Cancer (EORT QLQ-BR23). It contains 23 items, rated on a four-point scale ranging from 1 (not at all) to 4 (very much), assessing treatment side effects, arm symptoms, body image symptoms and sexual function. Scores range from 0 to 100 points.
Mood | Day 1
  It will be evaluated by means of the Spanish version of the Mood Evaluation Scale (EVEA). This questionnaire evaluates mood through 16 items, scored from 0 to 10 and divided into four categories (sadness-depression, anxiety, danger-hostility and happiness).
Kinesiophobia | Day 1
  It will be evaluated by means of the Spanish validation of the fear avoidance components scale (FACS-Sp). The questionnaire consists of 20 items evaluated on a 6-point Likert scale, where 0 indicates "strongly disagree" and 5 indicates "strongly agree". It has a maximum score of 100 points, with higher scores indicating more entrenched fear avoidance beliefs. Severity levels are classified as follows: subclinical (0-20), mild (21-40), moderate (41-60), severe (61-80) and extreme (81-100).
Anxiety and depression | Day 1
  It will be assessed using the Hospital Anxiety and Depression Scale (HADS). It consists of 14 items with two subscales, seven items assess anxiety and seven assess depression. The score of each subscale ranges from 0 to 21 points and a cut-off point equal to or higher than 11 points has been established to consider anxiety and depression states.

OTHER OUTCOMES:
Semi-structured interview, Perceived barriers | Day 1
  Qualitative variables will be collected through a semi-structured interview based on an interview guide. The interview will include questions that seek to know if the person performs physical exercise in breast cancer patients before, in process or after chemotherapy treatment, and the barriers they perceive to exercise. The interviews will be audio-recorded with the permission of the interviewees.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultat de Fisioteràpia Valncia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided